CLINICAL TRIAL: NCT06493487
Title: Integrated Neuromuscular Inhibition Technique Versus Instrument Assissted Soft Tissue Mobilization In Patients With Chronic Planter Fasciitis
Brief Title: INIT Versus IASTM In Patients With Chronic PF
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, esraa khairy afify esmail, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: INIT versus IASTM in PF
Record Dates: First submitted 2024-06-29; First posted 2024-07-10 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-06

CONDITIONS: Planter Fasciitis
Keywords: planter fasciitis; integrated neuromuscular inhibition technique (INIT); Instrument-Assisted Soft Tissue Mobilization (IASTM)

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- integrated neuromuscular inhibition technique (Experimental): integrated neuromuscular inhibition in addition to conventional treatment
  Interventions: Other: integrated neuromuscular inhibition technique
- instrument assisted soft tissue mobilization (Experimental): instrument assisted soft tissue mobilization technique (IASTM) in addition to conventional treatment
  Interventions: Other: instrument assissted soft tissue mobilization
- conventional treatment (Placebo Comparator): (home education program, therapeutic ultrasound, plantar fascia stretching, intrinsic muscle strengthening of foot, Self stretching of calf muscle using a towel and Ice Massage using frozen bottle).
  Interventions: Other: convential treatment

INTERVENTIONS:
Other: integrated neuromuscular inhibition technique — integrated neuromuscular inhibition technique for gastrocniemus muscle
  Arms: integrated neuromuscular inhibition technique
Other: instrument assissted soft tissue mobilization — instrument assissted soft tissue mobilization for calf muscle
  Arms: instrument assisted soft tissue mobilization
Other: convential treatment — convential treatment (home education program, therapeutic ultrasound, plantar fascia stretching, intrinsic muscle strengthening of foot, Self stretching of calf muscle using a towel and Ice Massage using frozen bottle).
  Arms: conventional treatment

SUMMARY:
1. To investigate integrated neuromuscular inhibition versus Instrument assisted soft tissue mobilization on general pain intensity in patient with chronic plantar fasciitis.
2. To investigate integrated neuromuscular inhibition versus Instrument assisted soft tissue mobilization on pain intensity at initial morning step in patient with chronic plantar fasciitis.
3. To investigate integrated neuromuscular inhibition versus Instrument assisted soft tissue mobilization on pain pressure threshold in patient with chronic plantar fasciitis.
4. To investigate integrated neuromuscular inhibition versus Instrument assisted soft tissue mobilization on active dorsiflexion ROM in patient with chronic plantar fasciitis.
5. To investigate integrated neuromuscular inhibition versus Instrument assisted soft tissue mobilization on functional disability in patient chronic plantar fasciitis.

5) Investigate integrated neuromuscular inhibition versus Instrument assisted soft tissue mobilization on functional disability in patient chronic plantar fasciitis.

DETAILED DESCRIPTION:
Plantar fasciitis (PF)is a degenerative syndrome of the plantar fascia resulting from repeated trauma at its origin on the calcaneus. Pain is generally caused by collagen degeneration at the origin of the plantar fascia at the medial tubercle of the calcaneus. It affects up to 10% of the general population. Functional risk factors include tightness in Gastrocnemius, soleus and weakness of intrinsic foot muscles because limited dorsiflexion of tight Achilles tendon strains the plantar fascia. Plantar fasciitis (PF), the most common cause of heel pain, it accounts for approximately 11% to 15% of foot symptoms presenting to physicians. The term plantar fasciitis implies an inflammatory condition. However, various lines of evidence indicate that this disorder is better classified as 'fasciosis' or 'fasciopathy' Plantar fasciitis. Main roles of plantar fascia are supporting longitudinal arch of the foot and providing shock absorption.if the tension on the plantar fascia exceeds the limits of the tissue, small tears can develop in the fascia. Repetitive tension and subsequent tearing can cause the fascia to become inflamed and painful. Plantar fasciitis is particularly common in runners, but is also noted among workers who stand for long periods.Any factor which is responsible for mechanical overloading of plantar fascia can be addressed as risk factors obesity, foot arch, decrease dorsiflexion ROM and tightness in calf muscles. One of the most common cause for limited ankle dorsiflexion range of motion (ADF)is gastrocnemius muscle tightness. The classic presentation of plantar fasciitis is pain on the sole of the foot at the inferior region of the heel. Pain is particularly bad with the first few steps taken on rising in the morning or after an extended refrain from weight-bearing activity. Often the pain diminishes after a few steps and through the course of the day, but returns if intense or prolonged weight bearing activity is carried out. Initially the heel pain may be diffuse or migratory; however, with time it usually focuses around the area of the medial tuberosity of calcaneum. Plantar heel pain is associated with impaired health-related quality of life including social isolation, a poor perception of health status and reduced functional capabilities.myofascial trigger points (MTrPs) in the calf muscle increase the stiffness and may reduce the dorsiflexion range of ankle joint which is one of the risk factor of plantar fasciitis.

Myofascial trigger points have the potential to create pain, limit ROM and restrict functional activities and should therefore be addressed as part of a comprehensive physical therapy program. Currently, a large variety of both manual and non-manual interventions exist for the deactivation of trigger points (TrPs). Manual approaches may include muscle energy techniques (METs), strain-counterstrain (SCS), myofascial release, proprioceptive neuromuscular facilitation, and ischemic compression.Integrated neuromuscular inhibition technique (INIT) is a method that includes three maneuvers in one. The three techniques are ischemic compression (IC) or trigger point release, strain counterstrain technique, and muscle energy technique (MET). In trigger point release, compression is given at the trigger point region and maintained for 15 seconds, while in strain counterstrain technique, the superficial fascia is stretched. MET works on the principle of reciprocal inhibition.Instrument-Assisted Soft Tissue Mobilization (IASTM) is uses specifically designed instruments to identify and treat myofascial restrictions. It is based off the principles of deep transverse friction massage. It is also known as Graston Technique. There are 6 stainless steel instruments which are specific for different regions and types of muscles which need to be targeted. It is designed to reduce fatigue of the clinician's hands and to detect lesions by amplifying the resonance felt through the instrument.

ELIGIBILITY:
Inclusion Criteria:

* Patient with history of plantar fasciitis more than three months ago.
* Plantar heel pain with first few steps upon walking in the morning and after prolonged rest.
* Patient's Age between 40-60 years old.
* Patient's Body mass index (BMI 18 to 29.9kg/m2).

Exclusion Criteria:

* Patients with any prior surgery to distal tibia, fibula, ankle joint or rear foot region.
* Presence of any red flags i.e., tumor, fracture, and heterotrophic ossification and had acute inflammatory condition at ankle-foot region were excluded from the study.
* Deformity of foot and ankle complex and subjects with referred pain due to sciatica and other neurological disorder.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
general pain intensity | change of general pain intensity through 4 weeks
  general pain intensity at planter aspect of foot will be measured by Visual analog scale (VAS): a horizontal line, 100 mm in length, anchored by word descriptors at each end (0 means no pain to 10 means worth pain). The VAS score is determined by measuring in millimeters from the left hand end of the line to the point that the patient marks.

SECONDARY OUTCOMES:
pain intensity in morning initial step | change of pain intensity in morning initial step through 4 weeks.
  pain intensity in morning initial step at planter aspect of foot will be measured by Visual analog scale (VAS): a horizontal line, 100 mm in length, anchored by word descriptors at each end.(0 means no pain to 10 means worse pain) The VAS score is determined by measuring in millimeters from the left hand end of the line to the point that the patient marks.

OTHER OUTCOMES:
Disability function of ankle joint | change of disability function of ankle joint through 4 weeks
  Disability function of ankle joint will be assisted by Arabic version of foot function index scale:
  The FFI (questionnaire) consists of 23 self-reported items divided into 3 subcategories on the basis of patient values: pain, disability and activity limitation. The patient has to score each question on a scale from 0 (no pain or difficulty) to 10 (worst pain imaginable or so difficult it requires help), that best describes their foot over the past week. The pain subcategory consists of 9 items and measures foot pain in different situations, such as walking barefoot versus walking with shoes. The disability subcategory consists of 9 items and measures difficulty performing various functional activities because of foot problems, such as difficulty climbing stairs. The activity limitation subcategory consists of 5 items and measures limitations in activities because of foot problems, such as staying in bed all day.
pain pressure threshold | change of pain pressure thershold through 4 weeks
  Pain pressure threshold will be measured by Pressure algometer (FPX 25 Wagner Instruments, Greenwich, CT, USA) was use for the measurement of PPT. Used to assess Pressure pain threshold (tenderness) over the lower medial trigger point in gastrocnemius muscle of the involved heel.
active ankle dorsiflexion range of motion | change of active ankle dorsiflexion range of motion through 4 weeks
  active ankle dorsiflexion range of motion will be measured by Electro goniometer:Used to measure active ankle dorsiflexion range of motion.

CONTACTS AND LOCATIONS:
Overall Officials: magda zahran, Ass.Prof, Study Director — faculty of physical therapy; Fatma Amin, Professor, Study Director — faculty of physical therapy; mohammed kaddah, professor, Study Director — Cairo University